CLINICAL TRIAL: NCT00679042
Title: Islet Transplantation in Type 1 Diabetic Patients Using the UIC Protocol, Phase 3
Brief Title: Islet Transplantation in Type 1 Diabetic Patients Using the University of Illinois at Chicago (UIC) Protocol
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CellTrans Inc. (Industry)
Responsible Party: Principal Investigator, Jose Oberholzer, Adjunct Professor of Surgery, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND11807-2007-0330
Expanded Access: NCT03791567 (Approved for marketing)
Record Dates: First submitted 2008-05-13; First posted 2008-05-16 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus Type 1; Type 1 Diabetes Mellitus; Islets of Langerhans Transplantation; Allogeneic Islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation; Basiliximab; Tacrolimus; Sirolimus; Etanercept; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): All subjects will receive up to 3 transplantations of allogeneic human islets of Langerhans.
  Interventions: Biological: Islets of Langerhans transplantation

INTERVENTIONS:
Biological: Islets of Langerhans transplantation — Each subject may receive 1-3 transplantations of allogeneic human islets of Langerhans and the following medications:
  Basiliximab 20 mg iv 2 hours before transplant and 20 mg iv 2 weeks post-transplant; Tacrolimus 1 mg p.o. bid adjusted to reach target trough levels of 3-6 ng/ml; Sirolimus 0.2 mg/kg loading dose, then 0.1 mg/kg p.o. daily adjusted to reach target trough levels of 10-15 ng/ml during the first 3 months post transplant and 7-10 ng/ml thereafter; Etanercept 50 mg iv 1 hour before transplant and 25 mg s.c. on days 3, 7,and 10 post-transplant; Exenatide 5-mcg s.c. bid for 1 week, then 10 mcg bid for 6 months after each transplant
  Other Names: Islets of Langerhan (Islets); Basiliximab (Simulect®); Tacrolimus (Prograf®); Sirolimus (Rapamune®); Etanercept(Enbrel®); Exenatide (Byetta®)

SUMMARY:
In an earlier Phase 1/2 clinical trial using the Edmonton Protocol of steroid free immunosuppression, investigators at University of Illinois at Chicago (UIC) demonstrated the safety of islet preparation, iset transplantation, and medical treatment at UIC. Therefore, the primary purpose of the present Phase 3 clinical trial is to demonstrate the safety and efficacy of allogeneic islet transplantation in improving glycemic control in Type 1 diabetic patients using the UIC protocol that was developed and proven effective during the Phase 1/2 clinical trial.

DETAILED DESCRIPTION:
This study is a Phase 3 single center, uncontrolled trial in which 1-3 allogeneic pancreatic islet transplants are performed for each study subject. Follow-up evaluations after transplant continue for 52 weeks after the final islet transplantation. Thereafter, subjects may enroll for a 5-year follow-up study and an additional 5 year to 10 year follow-up study to evaluate the function of the islets and to measure and regulate immunosuppressive drug levels and side effects.

The safety of islet transplantation depends primarily on the incidence of serious and unexpected complications or adverse events and the ability of the cell isolation laboratory to produce uncontaminated islet cell preparations with minimal endotoxin content.

All study subjects are followed for safety for one year. An independent Data Monitoring Committee (DMC), composed of 3 members who have training in medicine and/or organ transplantation, will review eligibility and safety data within 2 weeks after each islet transplantation and every two months thereafter. An independent monitor, who is knowledgeable about Good Clinical Practice (GCP) guidelines and regulations, monitors the study for compliance with 21 CFR and according to ICH GCP Guidelines. Within the Clinical Research Center, representatives of the Scientific Advisory Committee and the Research Subject Advocacy Program monitor safety. These entities report to the UIC Institutional Review Board (IRB), which also reviews safety data annually and on occurrence of serious adverse events. The principal investigator also reports serious adverse events to the US Food and Drug Administration (FDA).

Success: Islet transplantation is considered a success when subjects do not use insulin, and they achieve a fasting glucose level not exceeding 140 mg/dL more than three times in a week, and not exceeding two-hour post-prandial values of 180 mg/dL more than four times in a week.

Partial Success: Subjects who have a reduction in insulin requirements but who do not achieve insulin independence and present with a reduction in HbA1c and number of hypoglycemic episodes are considered to have partial success of islet transplantation. Reduction in insulin-requirements are assessed by comparing the pre-transplant insulin requirement recorded over two consecutive days (expressed as insulin units per kg) with the requirement on the two consecutive days preceding the subsequent islet infusion, and the requirements on two consecutive days at six months and again on two consecutive days at one year after the final transplant.

Failure: Absence of measurable levels of C-peptide after transplantation is considered as failure of islet cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for more than 5 years complicated by the following situations that persist despite intensive insulin management efforts:
* At least one episode of severe hypoglycemia in the past 3 years defined as an event with symptoms compatible with hypoglycemia in which the subject required the assistance of another person, and which was associated with either a blood glucose level <50 mg/dL (2.8 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration
* Reduced awareness of hypoglycemia, defined by the absence of adequate autonomic symptoms at capillary glucose levels of <54 mg/dL (3 mmol/l) as reported by the subject

Exclusion Criteria:

* Co-existing cardiac disease: myocardial infarction within the past 6 months, angiographic evidence of non-correctable coronary artery disease, ischemia on functional cardiac exam, heart failure
* Active alcohol or substance abuse, including cigarette smoking (must be abstinent for six months)
* Psychiatric disorder: schizophrenia, bipolar disorder, or major depression that is unstable on medication
* History of non-adherence to prescribed regimens
* Active infection including hepatitis C, hepatitis B, HIV
* TB by history, current infection, or under treatment for suspected TB
* History of malignancies except squamous or basal skin cancer
* Family history of MEN2 or MCT
* Stroke within the past 6 months
* BMI >27 kg/m2
* C-peptide response to glucagon stimulation, any C-peptide >0.3 ng/mL
* Inability to provide informed consent
* Age less than 18 or greater than 75 years
* Creatinine clearance <80 mL/min/1.73 m2 by 24-hour urine collection
* Serum creatinine consistently >1.5 mg/dL
* Macroalbuminuria >300 mg/24h
* Baseline Hb <12 gm/dL in women, <13 gm/dL in men
* Baseline liver function tests outside normal range
* Untreated proliferative retinopathy
* Positive pregnancy test, intent for pregnancy, male's intent to procreate, unwilling to use effective contraception, breast feeding
* Previous transplant or PRA reactivity >80%
* Insulin requirement >0.7 IU/kg/day
* HbA1c >12%
* Hyperlipidemia (fasting cholesterol >130 mg/dL or fasting triglycerides >200 mg/dL
* Medical condition requiring chronic use of steroids
* Use of Coumadin or other antiplatelet or anticoagulant therapy, or PT-INR >1.5
* Factor V deficiency
* Smoking tobacco
* Addison's disease
* Allergy to radiographic contrast material
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with medication absorption
* Treatment with antidiabetic medication other than insulin within 4 weeks of enrollment
* Use of any study medication within 4 weeks of enrollment
* Received live attenuated vaccine(s) within 2 months of enrollment
* Any medical condition that, in the opinion of the investigator, might interfere with safe participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-09-05 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2026-06-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Oberholzer, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Luu QF, Villareal CJ, Fritschi C, Monson RS, Oberholzer J, Danielson KK. Concerns and hopes of patients with type 1 diabetes prior to islet cell transplantation: A content analysis. J Diabetes Complications. 2018 Jul;32(7):677-681. doi: 10.1016/j.jdiacomp.2018.04.002. Epub 2018 Apr 17. PMID 29779835
- See also: The Chicago Diabetes Project Homepage — http://chicagodiabetesproject.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible patients with diabetes underwent a two-part screening phase to determine eligibility, followed by a waiting list period (as needed). The first subject consented on September 5, 2007. The last subject consented on November 4, 2014.
Pre-assignment Details: Potentially eligible patients with diabetes were to undergo a two-part screening phase to determine eligibility, followed by a waiting list period (as needed).
Groups:
- Treatment: All subjects will receive up to 3 transplantations of allogeneic human islets of Langerhans.
  Islets of Langerhans transplantation: Each subject may receive 1-3 transplantations of allogeneic human islets of Langerhans and the following medications:
  Basiliximab 20 mg iv 2 hours before transplant and 20 mg iv 2 weeks post-transplant; Tacrolimus 1 mg p.o. bid adjusted to reach target trough levels of 3-6 ng/ml; Sirolimus 0.2 mg/kg loading dose, then 0.1 mg/kg p.o. daily adjusted to reach target trough levels of 10-15 ng/ml during the first 3 months post transplant and 7-10 ng/ml thereafter; Etanercept 50 mg iv 1 hour before transplant and 25 mg s.c. on days 3, 7,and 10 post-transplant; Exenatide 5-mcg s.c. bid for 1 week, then 10 mcg bid for 6 months after each transplant
Period: Transplant + 1 Year Follow Up
Arm/Group | Treatment
Started | 21
Completed | 19
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: 5-Year Follow Up
Arm/Group | Treatment
Started | 19
Completed | 5
Not Completed | 14
Not completed — In follow-up (ongoing) | 6
Not completed — Death | 1
Not completed — Did not consent to continue into 10-year follow up | 7
Period: 10-Year Follow Up
Arm/Group | Treatment
Started | 5
Completed | 0
Not Completed | 5
Not completed — In follow-up (ongoing) | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] — Age at enrollment
  years | 47.0 [21 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
weight [Median (Full Range); unit: kg] | 63.8 [52.5 to 83.4]
height [Median (Full Range); unit: cm] | 165 [150.9 to 181.9]
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.4 (2)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: Safety endpoints: Incidence and severity of events related to islet infusion, immunosuppression, and islet preparations
Time Frame: From first islet transplant through one year after last transplant (maximum 3 infusions possible), an average of 1 year
Population: Intent to treat and as treated
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
Participants
  TEAE | 21
  Serious TEAE | 11
  TEAEs rated as severe or beyond | 16
  TEAEs leading to death or discontinuation | 0

2. Primary Outcome: Number of Subjects Reaching the Efficacy Goal
Description: A successful primary endpoint was defined as HbA1c ≤ 6.5% at the one-year follow-up visit and absence of severe hypoglycemic events (SHE) from Day 28 post-first transplant to 1 year after first and last transplant.
  The primary analysis was to estimate the true rate of the composite favorable outcome at 1 year following first and last transplant in patients in the ITT population.
Time Frame: One year after islet transplant
Population: Intent to treat/as treated
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
Participants
  Success at 1 yr post first transplant | 8
  Success at 1 yr post last transplant | 11

3. Secondary Outcome: Number of Patients Presenting With Insulin Independence at Day 365 Post First and Last Transplant
Description: Number of patients presenting with insulin independence, including:
  Absence of exogenous insulin injection reported at Day 365.
  * Fasting capillary glucose level not exceeding 140 mg/dL (7.8 mmol/L) more than 3 times in a week (based on measuring capillary glucose levels a minimum of 7 times in a 7-day period) at Day 365 ± 28 days.
  * Fasting plasma glucose level ≤ 126 mg/dL (7.0 mmol/L) at Day 365 ± 28 days (if the fasting plasma glucose level is > 126 mg/dL [7.0 mmol/L], it must have been confirmed in an additional 1 out of 2 measurements).
  * Two-hour post-prandial capillary glucose not exceeding 180 mg/dL (10.0 mmol/L) more than 1 out of every 7 times in a week (based on measuring capillary glucose levels a minimum of 7 times in a 7-day period) at Day 365 ± 28 days.
  * Evidence of endogenous insulin production defined as fasting or stimulated C-peptide levels ≥ 0.5 ng/mL (0.16 nmol/L) at Day 365 ± 28 days
Time Frame: 1 year after islet infusion
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 21
Participants
  First Tx Day 365 Absence of exogenous insulin | 10
  Last Tx Day 365 Absence of exogenous insulin | 12
  First Tx Day 365 Fasting capillary glucose in a week not exceeding 140 mg/dL more than 3X | 7
  Last Tx Day 365 Fasting capillary glucose in a week not exceeding 140 mg/dL more than 3X | 4
  First Tx Day 365 Fasting plasma glucose ≤126 mg/dL | 10
  Last Tx Day 365 Fasting plasma glucose ≤126 mg/dL | 11
  First Tx Day 365 Post-prandial capillary glucose in a week: Not exceeding 180 mg/dL more than 1X/7X | 5
  Last Tx Day 365 Post-prandial capillary glucose in a week: Not exceeding 180 mg/dL more than 1X/7X | 3
  First Tx Day 365 C-peptide (fasting or stimulated) ≥0.5 ng/mL | 10
  Last Tx Day 365 C-peptide (fasting or stimulated) ≥0.5 ng/mL | 10

4. Secondary Outcome: Hypoglycemic Episodes by HYPO Score
Description: Hypoglycemic episodes will be measured by the Ryan hypoglycemic (HYPO) Score derived from the number and severity of hypoglycemic episodes recorded throughout the follow-up phase from Day 28 to Day 365.
  (From Ryan et al., 2004) "A HYPO score was generated based on a combination of scores from the 4 weeks of readings and the patients' self-reported episodes over the previous year using the scoring system found in online appendix 2 (available at http://diabetes.diabetesjournals.org). The record sheets returned by the patients were analyzed for the number of episodes of glucose values recorded as <2.5 mmol/l and between 2.5 and 2.9 mmol/l. Points were awarded if symptoms were absent or were neuroglycopenic rather than autonomic... Thus the more severe the problem with hypoglycemia, the higher the score." A Ryan score ranges from 0 (no event) to a cumulative sum of episode points of total events reported during the 4 weeks then multiplied by 13 to provide a 1-year value.
Time Frame: One year after the last transplant
Population: ITT
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 21
score on a scale
  Baseline (pre-Tx): number analyzed (Participants) | 12
  Baseline (pre-Tx) | 266 [2 to 1638]
  First Tx Day 365: number analyzed (Participants) | 19
  First Tx Day 365 | 40.6 [0 to 1234]
  Last Tx Day 365: number analyzed (Participants) | 19
  Last Tx Day 365 | 18.7 [0 to 1234]

5. Secondary Outcome: Reduction in Hypoglycemic Severity Measured by %Reduction in HYPO Score
Description: %reduction in Ryan HYPO Score [%(baseline score - 1-year post transplant score)/baseline] at time of evaluation.
Time Frame: One year after the first and last transplant
Population: ITT
Measure: Mean (Full Range); unit: percentage of HYPO baseline
Arm/Group | Treatment
Number analyzed (Participants) | 21
percentage of HYPO baseline
  % Reduction from baseline to first tx day 365: number analyzed (Participants) | 11
  % Reduction from baseline to first tx day 365 | 66.1 [-300 to 100]
  % Reduction from baseline to last tx day 365: number analyzed (Participants) | 11
  % Reduction from baseline to last tx day 365 | 90.1 [-106 to 100]

ADVERSE EVENTS:
Time Frame: From first islet transplant through one year after last transplant (maximum 3 infusions possible), an average of 1 year.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=21)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Hypoglycaemia (Endocrine disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia legionella (Infections and infestations) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=21)
Vomiting (Gastrointestinal disorders) | 17 (23)
fatigue (General disorders) | 16 (17)
anemia (Blood and lymphatic system disorders) | 15 (28)
asthenia (General disorders) | 14 (16)
acne (Skin and subcutaneous tissue disorders) | 14 (18)
Headache (Nervous system disorders) | 12 (12)
Abnormal loss of weight (Metabolism and nutrition disorders) | 13 (17)
Transaminases increased (Investigations) | 10 (12)
diarrhea (Gastrointestinal disorders) | 13 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Leukopenia (Blood and lymphatic system disorders) | 6 (12)
Mouth ulceration (Gastrointestinal disorders) | 7 (10)
Stomatitis (Gastrointestinal disorders) | 8 (9)
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 7 (7)
Low density lipoprotein increased (Investigations) | 5 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (16)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (21)
Dizziness (Nervous system disorders) | 9 (9)
Tremor (Nervous system disorders) | 6 (7)
Insomnia (Psychiatric disorders) | 8 (8)
Pollakiuria (Renal and urinary disorders) | 6 (6)
Nocturia (Renal and urinary disorders) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-08-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT00679042/Prot_000.pdf
  • Statistical Analysis Plan (2014-08-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT00679042/SAP_001.pdf